CLINICAL TRIAL: NCT05265026
Title: Effect of Aerobic Exercise Training on Fat-fraction of the Liver in Patients With Chronic Hepatitis B and Hepatic Steatosis: a Randomised Controlled Intervention Trial. The Fit Liver Study
Brief Title: Aerobic Exercise Training in Patients With Chronic Hepatitis B and Hepatic Steatosis
Acronym: FitLiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Sofie Jespersen, Principal Investigator, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21034236
Record Dates: First submitted 2022-02-11; First posted 2022-03-03 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Hepatitis B, Chronic; Hepatic Steatosis
MeSH Terms: conditions — Hepatitis B, Chronic; Fatty Liver | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Arm (Experimental): Three high intensity interval exercise sessions per week of 40 minutes duration per session. Exercise will be performed on ergometerbikes.
  Interventions: Behavioral: High Intensity Interval Training
- No Intervention (No Intervention): No lifestyle changes

INTERVENTIONS:
Behavioral: High Intensity Interval Training — A training session consists of 40 minutes as follows: 4x4 minutes at > 85% of heart rate maximum (HRmax) alternated by 3x3 minutes active recovery at (50-70% of HRmax) and a 10-min-warm-up (60-79% of HRmax) and 5- minute cool-down at ~ warm up intensity. HRmax was determined during the VO2max test at baseline visit. Minutes spent in the different heart rate zones is monitored during the session (zone 1: 60-69%, zone 2: 70-74%, zone 3: 75-79%, zone 4: 80-84%, zone 5: >85% of HRmax).
  Arms: Exercise Intervention Arm

SUMMARY:
This study is a randomised, controlled, unblinded, clinical intervention trial consisting of 12 weeks of aerobic exercise training. Thirty persons with chronic hepatitis B (CHB) and hepatic steatosis are randomised to either aerobic exercise training (intervention group, n=15) or no intervention (control group, n=15). The study will investigate the effects of the exercise intervention on the liver and the hypothesis is that the exercise group will reduce the fat-fraction of the liver after the intervention.

DETAILED DESCRIPTION:
Primary aim: To investigate whether regular aerobic exercise training will decrease the fat-fraction of the liver in persons with CHB and hepatic steatosis shown by magnetic resonance imaging (MRI) by use of Iterative Decomposition of water and fat with Echo Asymmetry and Least squares estimation (IDEAL-IQ).

Secondary aim: To investigate the effects of aerobic exercise training on hepatokine secretion in persons with CHB and hepatic steatosis. Also, to investigate if regular physical exercise will improve lipid- and glucose metabolism, liver status, markers of inflammation, body composition, and blood pressure.

Study participants will undergo pre and post the interventioon: Clinical examination with ECG, blood pressure measurements, blood sampling, oral glucose tolerance test, a hormone infusion of somatostatin and glucagon, -increasing the glucagon/insulin ratio mimicking an acute exercise bout, measuring the effect on circulating hepatokines and cytokines, fibroscan, VO2-max test, DXA scan, AX3 activity monitoring, nail fold capillaryscopy, IQOLA SF-36 and IPAQ-SF questionnaire, 24H food intake registration, MRI scan of the liver and optional liver biopsy. 6 and 12 months follow-up is planned.

The exercise intervention will be randomised 1:1 with no stratification: The training program includes three weekly supervised training sessions of 40 minutes/session over 12 weeks. Participants are instructed not to change their lifestyles during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B defined by HBsAg positive >6 months
* Positive HBV-DNA
* Age >30
* Hepatic steatosis diagnosed by Controlled Attenuated Parameter (CAP) >250 assessed by Transient Elastography or by ultrasound defined hepatic steatosis

Exclusion Criteria:

* HIV, HCV, HDV-co infection
* Primary biliary cholangitis
* Wilsons Disease
* Autoimmune hepatitis
* Hepatocellular carcinoma
* Antiviral medication
* Steatogenic medication (systemic corticosteroids, amiodarone, tamoxifen, valproic acid, and methotrexate)
* Average alcohol intake >30 g for men and >20 g for women pr. day
* Contraindications for MRI scan
* Coronary artery disease contraindicating HIIT
* Unable to understand and read written information for participants written consent
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Fat-Fraction of the Liver | From baseline to follow-up at 12 weeks
  Hepatic fat-fraction measured by MRI with IDEAL-IQ (%)

SECONDARY OUTCOMES:
Fibroblast growth factor 21 (FGF21) secretion | From baseline to follow-up at 12 weeks
  FGF21 (ng/L) secretion during a hormone infusion of somatostatin and glucagon
Follistatin secretion | From baseline to follow-up at 12 weeks
  Follistatin (ng/L) secretion during a hormone infusion of somatostatin and glucagon
Growth/differentiation factor 15 (GDF15) secretion | From baseline to follow-up at 12 weeks
  GDF15 (ng/L) secretion during a hormone infusion of somatostatin and glucagon
Angiopoietin-like 4 (ANGPTL4) secretion | From baseline to follow-up at 12 weeks
  ANGPTL4 (μg/L) secretion during a hormone infusion of somatostatin and glucagon
C-reactive protein (CRP) secretion | From baseline to follow-up at 12 weeks
  CRP (mg/L) secretion during a hormone infusion of somatostatin and glucagon
Interferon-ϒ secretion | From baseline to follow-up at 12 weeks
  Interferon-ϒ (pg/mL) secretion during a hormone infusion of somatostatin and glucagon
Interleukin-10 secretion | From baseline to follow-up at 12 weeks
  Interleukin-10 (pg/mL) secretion during a hormone infusion of somatostatin and glucagon
Interleukin-8 secretion | From baseline to follow-up at 12 weeks
  Interleukin-8 (pg/mL) secretion during a hormone infusion of somatostatin and glucagon
Interleukin-6 secretion | From baseline to follow-up at 12 weeks
  Interleukin-6 (pg/mL) secretion during a hormone infusion of somatostatin and glucagon
Interleukin-1 secretion | From baseline to follow-up at 12 weeks
  Interleukin-1 (pg/mL) secretion during a hormone infusion of somatostatin and glucagon
TNFα secretion | From baseline to follow-up at 12 weeks
  TNFα (pg/mL) secretion during a hormone infusion of somatostatin and glucagon
Visceral fat | From baseline to follow-up at 12 weeks
  Visceral fat assessed by MRI (kg)
Total fat mass | From baseline to follow-up at 12 weeks
  Total fat mass assessed by DXA scan (kg)
Total free fat mass | From baseline to follow-up at 12 weeks
  Total free fat mass assessed by DXA scan (kg)
Total lean body mass | From baseline to follow-up at 12 weeks
  Total lean body mass assessed by DXA scan (kg)
Body weight | From baseline to follow-up at 12 weeks
  Body weight (kg)
Blood pressure measurements | From baseline to follow-up at 12 weeks
  Systolic blood pressure (mmHg) and diastolic blood pressure (mmHg)
Physical fitness (VO2max) | From baseline to follow-up at 12 weeks
  Physical fitness assessed by VO2max (mL/kg/min)
Total physical activity | From baseline, at 6 weeks to follow-up at 12 weeks
  Total physical activity assessed by activity monitor (hours, minutes)
Moderate and vigorous physical activity (MVPA) | From baseline, at 6 weeks to follow-up at 12 weeks
  Moderate and vigorous physical activity (MVPA) activity monitor (hours, minutes)
Sedentary time (SED) | From baseline, at 6 weeks to follow-up at 12 weeks
  Sedentary time (SED) activity monitor (hours, minutes)
Hepatitis B virus (DNA) | From baseline to follow-up at 12 weeks
  Hepatitis B virus (DNA) (IU/mL)
Oral glucose tolerance test | From baseline to follow-up at 12 weeks
  Oral glucose tolerance test (mmol/L)
Glycated haemoglobin type 1AC (HbA1c) | From baseline to follow-up at 12 weeks
  Glycated haemoglobin type 1AC (HbA1c) (mmol/mL)
Fasting glucose | From baseline to follow-up at 12 weeks
  Fasting glucose (mmol/L)
Fasting Insulin | From baseline to follow-up at 12 weeks
  Fasting Insulin (pmol/L)
Lipid measurements | From baseline to follow-up at 12 weeks
  Total cholesterol (mmol/L), total triglyceride (mmol/L), low density lipoprotein (LDL) (mmol/L), high density lipoprotein (HDL) (mmol/L)
Alanine transaminase (ALT) | From baseline to follow-up at 12 weeks
  Alanine transaminase (ALT) (U/L)
Aspartate transaminase (AST) | From baseline to follow-up at 12 weeks
  Aspartate transaminase (AST) (U/L)
Fibrosis-4 (FIB-4) | From baseline to follow-up at 12 weeks
  Fibrosis-4 (FIB-4)
International Normalised Ratio (INR) | From baseline to follow-up at 12 weeks
  International Normalised Ratio (INR)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Physical Activity Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be fully anonymized then the data can be shared.

REFERENCES:
- [Derived] Jespersen S, Plomgaard P, Madsbad S, Hansen AE, Bandholm T, Pedersen BK, Ritz C, Weis N, Krogh-Madsen R. Effect of aerobic exercise training on the fat fraction of the liver in persons with chronic hepatitis B and hepatic steatosis: Trial protocol for a randomized controlled intervention trial- The FitLiver study. Trials. 2023 Jun 13;24(1):398. doi: 10.1186/s13063-023-07385-y. PMID 37312098